CLINICAL TRIAL: NCT02478047
Title: Comparative Effect Study Between Distal-proximal Point Association and Local Distribution Point Association in Chemotherapy-induced Nausea and Vomiting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin University of Traditional Chinese Medicine (Other)
Collaborators: National Basic Research Program, China (Other)
Responsible Party: Principal Investigator, Yi Guo, the Dean of Acupuncture and Moxibustion College, Tianjin University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014CB543202-01
Record Dates: First submitted 2015-05-19; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-05

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: to Evaluate the Effectiveness of Acupucnture in the Management of Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — ramosetron; Tropisetron; Dexamethasone; Antiemetics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- only antiemetic (Active Comparator): The participants in the control group received standard antiemetic alone. Standard antiemetic for all groups is based on American Society of Clinical Oncology cClinical pPractice gGuideline. The 5-hydroxytryptamine-3 (5-HT3) antagonist (Ramosetron, Tropisetron) and dexamethasone are administered before the chemotherapy treatment.
  Interventions: Drug: only antiemetic (Ramosetron, Tropisetron and dexamethasone)
- Matching points ST36+CV12 (Experimental)
  Interventions: Other: Matching points ST36+CV12 plus antiemetic drug
- Matching points PC6+CV12 (Experimental)
  Interventions: Other: Matching points PC6+CV12 plus antiemetic drug
- Matching points CV3+CV12 (Experimental)
  Interventions: Other: Matching points CV13+CV12 plus antiemetic drug

INTERVENTIONS:
Drug: only antiemetic (Ramosetron, Tropisetron and dexamethasone) — The control group will receive standard antiemetic alone. Standard antiemetic for all groups is based on American Society of Clinical Oncology clinical practice guideline. 5-hydroxytryptamine-3 (5-HT3) antagonist (Ramosetron, Tropisetron) and dexamethasone are supplied from the first day of chemotherapy, and lasting for 3-5 days.And plus antiemetic drug as the comparator group.
  Arms: only antiemetic
Other: Matching points ST36+CV12 plus antiemetic drug — Choose both Zusanli(ST36) and Zhongwan point(CV12). Manipulating until achieving a "de Qi" sensation, then the needles are connected through a electro-acupuncture apparatus, the positive poles are linked to the needle, and the reference poles are located near the acupoint about 1cm with a paster. Frequency 10Hz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10mA. The operation lasts for 30 min. The treatment is scheduled to occur within 30min-60min before chemotherapy infusion for 4 days.And plus antiemetic drug as the comparator group.
  Arms: Matching points ST36+CV12
Other: Matching points PC6+CV12 plus antiemetic drug — Choose both Neiguan(PC6) and Zhongwan point(CV12). Manipulating until achieving a "de Qi" sensation, then the needles are connected through a electro-acupuncture apparatus, the positive poles are linked to the needle, and the reference poles are located near the acupoint about 1cm with a paster. Frequency 10Hz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10mA. The operation lasts for 30 min. The treatment is scheduled to occur within 30min-60min before chemotherapy infusion for 4 days.And plus antiemetic drug as the comparator group.
  Arms: Matching points PC6+CV12
Other: Matching points CV13+CV12 plus antiemetic drug — Choose both Shangwan(CV13) and Zhongwan point(CV12). Manipulating until achieving a "de Qi" sensation, then the needles are connected through a electro-acupuncture apparatus, the positive poles are linked to the needle, and the reference poles are located near the acupoint about 1cm with a paster. Frequency 10Hz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10mA. The operation lasts for 30 min. The treatment is scheduled to occur within 30min-60min before chemotherapy infusion for 4 days.And plus antiemetic drug as the comparator group.
  Arms: Matching points CV3+CV12

SUMMARY:
The purpose of this study is to clarify whether distal-proximal point association is more effective than partial match point association by electro-acupuncture in the management of chemotherapy-induced nausea and vomiting .

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed as cancer and need to accept chemotherapy.
2. The score of Karnofsky ≥70
3. Patients of either gender and older than 18 years
4. Patients receiving chemotherapy both outpatients and inpatients
5. Patients receiving chemotherapy either the first or multiple cycle, but the patient will be taken in only one time
6. To receive chemotherapy containing cisplatin(DDP≥75mg/m2) or joint chemotherapy programmes of Anthracyclines(Adriamycin≥40mg/m2 or epirubicin≥60mg/m2)
7. Life expectancy≥ 6 months
8. Willing to participate in the study and be randomized into one of the four study groups.

Exclusion Criteria:

1. To receive radiotherapy and chemotherapy
2. Gastrointestinal tumors
3. Patients with serious liver disease or abnormal hepatorenal function (AST,ACT, and TBIL are 3 times more than normal, BUN and Cr are 2 times more than normal)
4. Presence of cardiac pacemaker
5. Active skin infection
6. Nausea and/or vomiting resulting from opioids or metabolic imbalance (electrolyte disturbances)
7. Patients unable to provide self-care or communication
8. Nausea and/or vomiting resulting from mechanical risk factors (i.e., intestinal obstruction)
9. Brain metastases
10. Women in pregnant and lactating period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
the frequency of Nausea and Vomiting | 3 weeks
the extent of Nausea and Vomiting | 3 weeks
Rhodes Index of Nausea, Vomiting and Retching | 3 weeks

SECONDARY OUTCOMES:
the condition of constipation and diarrhea | 3 weeks
gastric electrical activity (electrogastrogram) | 3 weeks
the life quality of the patients | 3 weeks
the Anxiety and Depression of the patients | 3 weeks

OTHER OUTCOMES:
the number of blood cells | 3 weeks
  the number of WBC,RBC,hemoglobin,PLT,the percents of GRA,LYM
cardial electrical activity | 3 weeks
hepatic function | 3 weeks
  The Outcome Measures will be assessed by blood, the metrics of ALT,AST,TBIL is IU/L,IU/L,and μmol/L.
other adverse effect during the chemotherapy | 3 weeks
renal function | 3 weeks
  The Outcome Measures will be assessed by blood, the metrics of BUN,Scr is mmol/L and μmol/L.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin University of TCM, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Gao L, Chen B, Zhang Q, Zhao T, Li B, Sha T, Zou J, Guo Y, Pan X, Guo Y. Acupuncture with different acupoint combinations for chemotherapy-induced nausea and vomiting: study protocol for a randomized controlled trial. BMC Complement Altern Med. 2016 Nov 8;16(1):441. doi: 10.1186/s12906-016-1425-1. PMID 27821107